CLINICAL TRIAL: NCT04748744
Title: Value of Butyrylcholinesterase as a Marker of Surgical Site Infection Following Surgery for Colorectal Diseases
Status: Completed | Type: Observational
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Francesk Mulita, Principal Investigator, University Hospital of Patras
Other Study IDs: 4025
Record Dates: First submitted 2020-11-03; First posted 2021-02-10 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Disorders; Colorectal Neoplasms
Keywords: butyrylcholinesterase
MeSH Terms: conditions — Colorectal Neoplasms; Butyrylcholinesterase deficiency | interventions — Butyrylcholinesterase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing colorectal surgery
  Interventions: Combination Product: Butyrylcholinesterase

INTERVENTIONS:
Combination Product: Butyrylcholinesterase — Value of Butyrylcholinesterase as a Marker of Surgical Site Infection Following Surgery for Colorectal Diseases

SUMMARY:
Butyrylcholinesterase (BChE) is an α-glycoprotein synthesized in the liver. BchE's serum level decreases in many clinical conditions such as acute and chronic liver damage, inflammation, injury and infections, and malnutrition. The Investigators prospectively evaluate patients undergoing elective procedures for colorectal diseases. Blood samples are collected preoperatively (at day 0), post-operatively in the recovery room (day 1), and on the subsequent four days (days 2, 3, 4, and 5) for assessment of BChE, C-reactive protein, and white blood cell concentrations. The same surgical team operates all patients and is blinded to the study. Patients are monitored for post-operative infection by using standard laboratory and clinical methods. If surgical site infection (SSI) is suspected the wound is swabbed and empirical antibiotics are started. The aim of the current trial is to study whether BChE is a reliable marker for the presence of SSI in patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
Butyrylcholinesterase (BChE or BuChE) is a cholinesterase enzyme that is very similar to acetylcholinesterase (AChE). However, though the role and function of AChE in the human body are widely studied and known, BChE is usually referred to as an 'orphan enzyme' because its specific physiological role is still under question. Lastly, it has been found, however, that BChE has more specific functions than it was previously believed and acetylcholine (ACh), which will be further analyzed, can affect the immune system and is associated with inflammation-related events. Butyrylcholinesterase is an enzyme that for several years was not considered to have a specific physiological role but lately, it has been observed that plays an important role in inflammation as acetylcholine is a major player of the 'cholinergic anti-inflammatory pathway' inhibiting inflammation. It has been proved that BChE activity can be affected by several diseases. Low-grade inflammation is associated with an increase of its levels whereas a reduction is observed when systemic inflammation is present. However, future research is needed in order to be widely used in clinical practice as a biomarker for several pathological conditions involving inflammation. Therefore, the aim of this study is to present information about butyrylcholinesterase, its function, and its role in the human body, highlighting its association with inflammation analyzing past studies about this subject. The Investigators prospectively evaluate patients undergoing elective procedures for colorectal diseases. Blood samples are collected preoperatively (at day 0), post-operatively in the recovery room (day 1), and on the subsequent four days (days 2, 3, 4, and 5) for assessment of BChE, C-reactive protein, and white blood cell concentrations. The same surgical team operates all patients and is blinded to the study. Patients are monitored for post-operative infection by using standard laboratory and clinical methods. If surgical site infection (SSI) is suspected the wound is swabbed and empirical antibiotics are started. The aim of the current trial is to study whether BChE is a reliable marker for the presence of SSI in patients undergoing colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Operation for colorectal disease
* Older than 18 years old

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical Site Infection in patients older than 18 years old that will have an operation for colorectal disease
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Value of Butyrylcholinesterase as a Marker of Surgical Site Infection Following Surgery for Colorectal Diseases | November 6th 2019 to March 1st 2023
  Blood samples will be collected preoperatively by the investigators (at day 0), post-operatively in the recovery room (day 1), and on the subsequent four days (days 2, 3, 4, and 5) for assessment of serum BChE. The normal range of this BchE in our laboratory is 2.8-7.4 KU/L

CONTACTS AND LOCATIONS:
Locations (1):
- Francesk Mulita, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Panos G, Mulita F, Akinosoglou K, Liolis E, Kaplanis C, Tchabashvili L, Vailas M, Maroulis I. Risk of surgical site infections after colorectal surgery and the most frequent pathogens isolated: a prospective single-centre observational study. Med Glas (Zenica). 2021 Aug 1;18(2):438-443. doi: 10.17392/1348-21. PMID 34080408
- [Result] Mulita F, Liolis E, Akinosoglou K, Tchabashvili L, Maroulis I, Kaplanis C, Vailas M, Panos G. Postoperative sepsis after colorectal surgery: a prospective single-center observational study and review of the literature. Prz Gastroenterol. 2022;17(1):47-51. doi: 10.5114/pg.2021.106083. Epub 2021 May 23. PMID 35371356